CLINICAL TRIAL: NCT06683859
Title: Critical Anatomical Variants in Preoperative Computed Tomography of Paranasal Sinuses and Nasal Cavity : a Study in a Tertiary Care Center of Nepal
Brief Title: Variants of Paranasal Sinuses in Nepali Population
Status: Completed | Type: Observational
Sponsor: Grande International Hospital, Nepal (Other)
Responsible Party: Principal Investigator, PRAJWAL DAHAL, Consultant Radiologist, Grande International Hospital, Nepal
Other Study IDs: 17/2023
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Paranasal Sinuses
Keywords: Computed Tomography (CT); Paranasal Sinuses (PNS); Functional Endoscopic Sinus Surgery(FESS)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paranasal sinus of patients with no obvious pathology

SUMMARY:
The variants of paranasal sinuses (PNS)and nasal cavity are of clinical importance since some variants are susceptible to recurrent infection. Moreover, during functional endoscopic sinus surgery, knowledge of anatomy is of utmost importance in order to prevent injury of vital structures like optic nerves, carotid arteries etc. However, there is lack of study enrolling adequate number of patients in our country. Critical variants are often underreported by radiologists. Thus, it is imperative to know true prevalence of different anatomical variants.

DETAILED DESCRIPTION:
The nasal cavity and paranasal sinuses(PNS) together constitute single anatomical and functional unit. There are different anatomical variants of paranasal sinuses and nasal cavity. This is the anatomical structure with most variation and computed tomography(CT) is frequently done to evaluate anatomy of PNS and nasal cavity. Knowledge of anatomical variants is important for early diagnosis of pathology in the region and to prevent complications during functional endoscopic sinus surgery(FESS). Different anatomical variants frequently seen in CT of PNS and nasal cavity include deviated nasal septum, bony spur, concha bullosa, paradoxical nasal turbinate, agger nasi cells, bulla ethmoidalis, haller cells, onodi cells, different degree of pneumatization of sphenoid sinus etc. Anatomical variation of these structures differs in different ethnic groups. Some variants like onodi cells, complete sellar pneumatization of sphenoid sinus, anterior ethmoid artery traversing ethmoid air cells, dehiscent optic nerve and carotid artery pose structure around them into risk during surgery. If exact prevalence of these anatomical variations is known, it becomes easy for surgeons to approach lesions in the area easily. Some variants like haller cells, ager nasi cells, bulla ethmoidalis block osteomeatal complex and drainage pathway of frontal sinuses. Sinusitis may be refractory to medications due to these variants. We could find three studies done in our country and the sample size ranges from 76 to 218. We are aiming for larger study which could provide more accurate picture of prevalence of different anatomical variants. CT of PNS is done frequently in our hospital and we rarely collect data from the images for research purpose. There would be utilization of those data as well. Patient need not pay extra or receive extra radiation for the study. We think the study is very noble and would be a great help for surgeons and clinicians in the country.

ELIGIBILITY:
Inclusion Criteria:

* CT scan of PNS of patients > 13 years referred for various reasons.
* CT scan of Head referred to our department for various reasons.

Exclusion Criteria:

* CT of PNS and head done for evaluation of trauma and tumors
* CT of Patients age less than 13 years .

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nepali Population
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of Anatomical variants of paranasal sinuses in Nepali population | 6 months
  Prevalence of agger nasi cell, haller cell, different types of olfactory fossa

CONTACTS AND LOCATIONS:
Locations (1):
- Tokha Road, Dhapasi, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
I, the principal investigator choose not to share the plan

REFERENCES:
- [Background] Shrestha KK, Acharya K, Joshi RR, Maharjan S, Adhikari D. Anatomical Variations of the Paranasal Sinuses and the Nasal Cavity. Nepal Med Coll J. 2019 Mar 31;21(1):7-11